CLINICAL TRIAL: NCT05961540
Title: Study on the Construction and Application of Breastfeeding Behavior Intervention Program for Mothers of Infants With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHFudan
Record Dates: First submitted 2023-06-07; First posted 2023-07-27 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Heart Defects, Congenital; Breast Feeding
Keywords: Heart Defects, Congenital; Breast Feeding; Infant, Newborn; Feeding intervention
MeSH Terms: conditions — Heart Defects, Congenital; Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care group (Other): The management of infants with CHD and their mothers is based on the current breastfeeding process and care protocols at the Cardiovascular Centre of the Children's Hospital of Fudan University.
  Interventions: Other: Conventional care
- Breastfeeding intervention program (Experimental): Implement intervention programs to improve breastfeeding behaviour among mothers of infants with CHD and observe ongoing changes.
  Interventions: Behavioral: Breastfeeding behavioural intervention for mothers of infants with CHD

INTERVENTIONS:
Other: Conventional care — 1. Instruct parents to follow up with the baby at the doctor's appointment.
  2. Provide telephone follow-up visits at 1 month, 3 months, and 6 months of age to assess the baby's feeding and physical development (height and weight).
  Arms: Conventional care group
Behavioral: Breastfeeding behavioural intervention for mothers of infants with CHD — Based on the Behavioural Change Wheel theory,the intervention program is developed and implemented to promote the change in breastfeeding behavior of mothers with CHD infants,so as to improve the exclusive breastfeeding rate of this population.Specific programs include:
  1. Evaluate signs of hunger and satiety in infants.
  2. Family visits, face-to-face guidance on breastfeeding skills, breast milk storage and management.
  3. Training methods for promoting breast milk secretion.
  4. To explain common feeding difficulties manifestations and treatment methods in infants with CHD.
  5. Establish a breastfeeding promotion alliance.
  6. Teach mothers to weigh their babies before and after breastfeeding to determine breast milk intake.
  7. Assess and guide the growth and development of infants with CHD.
  Arms: Breastfeeding intervention program

SUMMARY:
This study is a randomized block trial designed to evaluate the effectiveness of a breastfeeding behavioural intervention program for mothers of infants with congenital heart disease (CHD). The purpose of this study is to compare exclusive breastfeeding rates, changes in weight-for-age z-scores (ΔWAZ) and height-for-age z-scores (ΔHAZ), and maternal breastfeeding behaviour between the intervention group and the control group at 1, 3, and 6 months of age.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) refers to an abnormality in the development of the heart and major blood vessels during fetal development. The prevalence of CHD in China is 8.94 per 1,000 live births and poses a significant public health concern for children's well-being. Infants with CHD often suffer from fluid restriction, nausea, belching, choking and stuttering due to structural changes in the heart and abnormal haemodynamics, which pose a challenge to their nutritional intake. The World Health Organization (WHO) advises that breastfeeding is the best way to nourish infants. Breastfeeding should begin within one hour of birth, and exclusive breastfeeding means that no other food or liquid, including water, should be continued for the first six months of life. The Expert Consensus on Nutritional Support for Children with Congenital Heart Disease recommends breast milk as the optimal nutrition for newborns and encourages infants with CHD to breastfeed. While breastfeeding offers benefits such as immune system enhancement, improved nervous system development, and increased intelligence for infants with CHD, breastfeeding rates are low in this population and interruptions are frequent. A behaviour change program based on the behaviour change wheel will be implemented at the Children's Hospital of Fudan University to enhance breastfeeding behaviour in mothers of infants with CHD, with the aim of increasing the rate of exclusive breastfeeding in this population.

ELIGIBILITY:
Inclusion Criteria:

* For infants

CHD was diagnosed within 14 days of birth.

From birth to 14 days old.

Exclusive breastfeeding or mixed feeding during enrollment.

* For mothers

The mother is the primary caretaker for the infant with CHD.

The mother has a smartphone and has the skills to use it.

She has good reading and communication skills and can work fully with others.

In good physical health with no clear disability, such as severe cardiovascular disease, etc.

In good mental health, without any clearly diagnosed anxiety disorders, depression, etc.

Mothers must be at least 18 years old.

Exclusion Criteria:

* For infants

Congenital anomalies such as gastrointestinal anomalies, facial anomalies, cleft lip and palate, and various syndromes due to chromosomal abnormalities are combined.

Cardiac surgery was performed within 14 days of birth.

The infant is not breastfed according to medical standards (for example, with galactosemia, phenylketonuria, or maple glycosuria).

* For mothers

Mothers with mental illness, cognitive impairment, etc. who struggle to communicate effectively.

Those who have contraindications to breastfeeding, such as long-term use of specific types of drugs such as chemotherapy drugs, opioids, anti-epileptic drugs, anti-depressants, psychotropic drugs, etc.

Systemic infectious diseases during feeding include HIV positive, active or untreated tuberculosis, recent syphilis infection, etc.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding rate | At the age of 1month
  The exclusive breastfeeding rate equals (the number of CHD infants who choose exclusive breastfeeding) divided by (the total number of CHD infants) multiplied by 100%.
Exclusive breastfeeding rate | At the age of 3 months
  The exclusive breastfeeding rate equals (the number of CHD infants who choose exclusive breastfeeding) divided by (the total number of CHD infants) multiplied by 100%.
Exclusive breastfeeding rate | At the age of 6 months
  The exclusive breastfeeding rate equals (the number of CHD infants who choose exclusive breastfeeding) divided by (the total number of CHD infants) multiplied by 100%.

SECONDARY OUTCOMES:
Breastfeeding Behavior Questionnaire for Mothers of Infants with CHD | At baseline and at 6 months of age.
  This questionnaire was created by us with a total of 21 items, which include five dimensions of breastfeeding behavior of mothers of CHD infants: mothers' attention to breastfeeding of children with congenital heart disease, identification of signals of hunger and satiety of infants, breastfeeding skills, methods to promote lactation, and identification and treatment of choking milk during breastfeeding of CHD infants. The questionnaire uses the Likert5-level scoring method, with a score of 0-105. The higher the score, the better the breastfeeding behavior of CHD infant mothers.
ΔWAZ at 1 month of age compared to birth, separated into two groups. | At the age of 1month
  The infant's family has created their own digital scale that is as precise as the one used in the hospital. The weight measurement is accurate to 0.01 kilograms. For accurate measurement, it is recommended to weigh the baby at the age of one month in the early morning. Before measuring, the baby scale should be reset to zero, and the baby should be undressed in clothes and diapers. The baby's weight will be converted to WAZ. The WAZ at the age of 1 month minus the WAZ converted from birth weight is the ΔWAZ at the age of 1 month after birth.
ΔWAZ at 3 months of age compared to birth, separated into two groups. | At the age of 3 months
  The infant's family has created their own digital scale that is as precise as the one used in the hospital. The weight measurement is accurate to 0.01 kilograms. For accurate measurement, it is recommended to weigh the baby at 3 months of age in the early morning. Before measuring, the baby scale should be reset to zero, and the baby should be undressed in clothes and diapers. The baby's weight will be converted to WAZ. The WAZ at the age of 3 months minus the WAZ converted from birth weight is the ΔWAZ at the age of 3 months after birth.
ΔWAZ at 6 months of age compared to birth, separated into two groups. | At the age of 6 months
  The infant's family has created their own digital scale that is as precise as the one used in the hospital. The weight measurement is accurate to 0.01 kilograms. For accurate measurement, it is recommended to weigh the baby at 6 months of age in the early morning. Before measuring, the baby scale should be reset to zero, and the baby should be undressed in clothes and diapers. The baby's weight will be converted to WAZ. The WAZ at the age of 6 months minus the WAZ converted from birth weight is the ΔWAZ at the age of 6 months after birth.
ΔHAZ at 1 month of age compared to birth, separated into two groups. | At the age of 1 month
  The baby's family has prepared a height measuring tool that is as precise as the ones used in hospitals. The height measurement is within 0.1 centimeter accuracy. The baby's height should be measured early in the morning on the day when the baby is 1 month old. The baby's length will be converted into a HAZ. The HAZ at the age of 1 month minus the HAZ converted from birth length is the ΔHAZ at the age of 1 month after birth.
ΔHAZ at 3 months of age compared to birth, separated into two groups. | At the age of 3 months
  The baby's family has prepared a height measurement tool that is as precise as those used in hospitals. The height measurement is within 0.1 centimeter accuracy. The baby's height should be measured early in the morning on the day the baby is 3 months old. The baby's length will be converted into a HAZ. The HAZ at the age of 3 months minus the HAZ converted from birth length is the ΔHAZ at the age of 3 months after birth.
ΔHAZ at 6 months of age compared to birth, separated into two groups. | At the age of 6 months
  The baby's family has prepared a height measurement tool that is as precise as those used in hospitals. The height measurement is within 0.1 centimeter accuracy. The baby's height should be measured early in the morning on the day the baby is 6 months old. The baby's length will be converted into a HAZ. The HAZ at the age of 6 months minus the HAZ converted from birth length is the ΔHAZ at the age of 6 months after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gu, Doctor, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China